CLINICAL TRIAL: NCT03754725
Title: A Phase 1/2a Exploratory Clinical Trial to Evaluate the Safety of Oral Deferiprone (14 Days) Including Its Effect on Decreasing the Content of Iron in Subjects With Aneurysmal Subarachnoid Hemorrhage (aSAH) sIRB
Brief Title: Ferritin and Iron Burden in SAH sIRB
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00110138
Record Dates: First submitted 2018-11-24; First posted 2018-11-27 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: SAH; Dementia
Keywords: Deferiprone
MeSH Terms: conditions — Dementia | interventions — Deferiprone; Ferritins; Mental Status and Dementia Tests

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deferiprone (Experimental): This is the drug arm (deferiprone). Patients will receive oral deferiprone
  Interventions: Drug: Deferiprone pill; Behavioral: Montreal Cognitive Assessment
- Control (Placebo Comparator): this group will only receive the placebo (sugar pill)
  Interventions: Drug: placebo; Behavioral: Montreal Cognitive Assessment

INTERVENTIONS:
Drug: Deferiprone pill — 1000 mg of deferiprone (oral) BID (15 mg/Kg)
  Other Names: Ferritin
  Arms: Deferiprone
Drug: placebo — patients will receive placebo orally
  Arms: Control
Behavioral: Montreal Cognitive Assessment — Neurocognitive assessment, lower score indicates lower cognitive level
  Other Names: MoCA

SUMMARY:
Ruptured cerebral aneurysms lead to subarachnoid hemorrhage (SAH),that has a high morbidity and mortality rate, the severity of which is predicted by the "Hunt-Hess grade" (HHG).

SAH leads to iron (Fe) and hemoglobin (Hb) accumulation in the brain, which is toxic for neurons. Ferritin (iron reported in the brian) and iron overload leads to brain atrophy, specifically in the mesial temporal lobe (hippocampus, impairing patients' cognition. It is estimated that 50% of survivors have cognitive deficits.

Most of the survivors of SAH could not return to work. Iron chelation therapy has been recently gaining ground as a therapeutic intervention in intraparenchymal hemorrhage and in SAH. However, there has not been any study that assess the iron deposition in the brain and the level of ferritin in the cerebrospinal fluid of SAH patients. The investigators propose to conduct a randomized trial using Deferiprone (oral chelating agent, "De") + standard of care versus standard of care in patient with SAH to:

1. assess the level of ferritin (Ft) in CSF (CSF withdrawn from ventriculostomy tube),
2. assess functional outcomes measured by the Montreal Cognitive Assessment (MoCA) score, a score used to assess the level of dementia, mainly in Alzheimer disease patients.
3. quantify the the total iron deposition in the brain based on MRI

DETAILED DESCRIPTION:
I) SIGNIFICANCE

1) Significance and Incidence and Burden of the disease Intracranial aneurysm is a prevalent disease estimated around 2-5% of the population. Aneurysm rupture leads to aneurysmal subarachnoid hemorrhage , which have a tremendous impact on the patient's health, and a high mortality rate (~60%), with a large proportion of the survivors becoming functionally dependent. It accounts for 27% of all stroke-related years of life lost before age 65, and it has a predilection for a relatively younger age. Survivors have long term cognitive deficits and memory impairment in their productive years with major responsibilities with respect to work and family. Despite that, only one-third have neurological deficits. Most of the survivors could not return to work. Poor functional outcomes are related to iron and heme toxicity with resultant delayed cerebral ischemia , early brain injury , hydrocephalus and cerebral edema. As of today, there has not been any intervention that improves neurocognitive outcomes in these patients. The investigators postulate that iron chelation therapy can decrease the amount of Iron (Fe) deposition in the brain, reduce ferritin (Ft) in patients' cerebrospinal fluid (CSF) and potentially improve functional outcome.

Our group was the first in the world to detect and quantify Fe concentration at the interface of brain aneurysms' wall and brain tissue using QSM-MRI sequence. This technique allowed us to detect microbleeds associated with sentinel headache in subjects with IAs and negative non-contrast head CT and negative lumbar puncture. In this proposal, the investigators will also use high-resolution MRI sequence to assess difference in volumes of amygdala and hippocampus and correlate that with CSF-ferritin.

This will make our proposal the first go/no-go randomized double-blind placebo vs. deferiprone trial that attempts to establish Ft (a reporter of total Fe in the brain and CSF) as a biomarker of neurocognitive decline specifically in subarachnoid hemorrhage subjects and test the effect of deferiprone in decreasing the levels of Ft and therefore ameliorate the neurocognitive decline associated with this disease. If our hypothesis is validated, then this would set the stage for a phase 3 clinical trial and test our hypothesis in larger cohort of subjects.

III) PRELIMINARY DATA (obtained with collaboration with our colleagues in Europe):

To provide proof-of-concept of the effect of deferiprone on the levels of Ft in the CSF of subjects with aneurysmal subarachnoid hemorrhage (aSAH), Tthe investigators conducted a pilot study to analyze the concentration Ft in the CSF of subjects with aSAH and Hunt and Hess grade 1-3. Fourteen subjects were included (7 with only cisternal SAH but no intraventricular hemorrhage (IVH), and 7 subjects with cisternal aSAH and IVH). Their CSF (2-3 cc) were drawn daily (from day 0 to day14) and analyzed with Fe-ELISA kit. Then 4 subjects (2 with aSAH without IVH and 2 with SAH and IVH) were treated with 1000 mg of deferiprone twice orally for 14 days. The mean Ft level in subjects with aSAH without IVH was 900ng/ml vs. 420 ng/ml for those receiving deferiprone. The mean Ft level of patients with SAH and IVH was 1500ng/ml compared to 690 ng/ml in the deferiprone group. This small pilot study provided proof-of-concept that 1) aSAH increases the CSF-Ft in human, and this effect can be reduced significantly with deferiprone, and 2) aSAH associated with IVH increases furthermore CSF-Ft, which is also reduced significantly by deferiprone.

ELIGIBILITY:
Inclusion criteria:

1. Age greater than or equal to 18 and less than or equal to 75 years.
2. Historical modified Rankin Scale Score (mRS) 0-1 (pre-subarachnoid hemorrhage onset).
3. World Federation of Neurosurgical Societies SAH Scale (WFNS) grade less than or equal to 4, due to a spontaneous SAH attributed to a ruptured cerebral aneurysm. Initial WFNS grade may be determined at admission or enrollment, preferably after the patient's mental status has been optimized by resuscitation and interval treatment of hydrocephalus (i.e., placement of intraventricular catheter or lumbar puncture [LP]) or reversal/wearing-off of sedating medications used commonly during patient transfers and transport or procedure related anesthesia.
4. Admission head CT showing modified Fisher grade 1-4 due to aneurysmal subarachnoid hemorrhage (aSAH) primarily in the supratentorial space. The Modified Fisher CT rating scale is: Grade 1 (minimal or diffuse thing SAH without intraventricular hemorrhage); Grade 2 (minimal or thin SAH with intraventricular hemorrhage), Grade 3 (thick cisternal clot without intraventricular hemorrhage), Grade 4 (thick cisternal clot with intraventricular hemorrhage).
5. Location and pattern of the SAH must have the majority of the SAH in the supratentorial space caused by either an intradural anterior circulation aneurysm or a basilar apex/posterior circulation aneurysm with primarily supratentorial hemorrhage extension. Angiographic location of the aneurysm will be confirmed by catheter digital subtraction angiography usually obtained during the coil embolization procedure.
6. Onset of symptoms of aSAH (ictus) occurred < 24 hours prior to presentation at the treating facility.
7. Initiation of aneurysm securement procedure occurred < 48 hours from the ictus and less than 12 hours from admission to the treating facility.
8. All aneurysm(s) suspected to be responsible for the hemorrhage or potentially responsible for the hemorrhage must be secured in the following manner prior to enrollment: endovascular Coil Embolization with a post-embolization Raymond-Roy Score of 1 (Complete) or 2 (Residual Neck).
9. Ability to screen the patient and obtain head CT and CT perfusion on admission and follow after recovering from anesthesia following the aneurysm coiling procedure, the patient must remain a WFNS SAH grade less than or equal to 4 without evidence of a significant new focal neurological deficit including monoparesis / monoplegia, hemiparesis / hemiplegia, or receptive, expressive or global aphasia. New minor cranial nerve defect without any other new findings is permissible. If a national institute of health stroke scale (NIHSS) score was obtained prior to the aneurysm coiling procedure, a post-coiling (pre-enrollment) NIHSS score must not have increased by 4 points or more and Glasgow coma score must not be decreased by 2 points or less. The clinician should use their best clinical judgment as to whether a significant neurological decline has occurred due to the coiling procedure.
10. Ability to obtain MRI for ischemic changes evaluation.
11. Subject's Legally Authorized Representative (LAR) has provided written informed consent.

Exclusion Criteria:

1. Angio-negative SAH.
2. A likely hemorrhage event within several days prior to admission related hemorrhage ictus due to the increased risk of early vasospasm.
3. Prior sentinel headache with negative CT or prior sentinel headache where the patient did not seek medical attention does not exclude the patient.
4. Surgical clipping of the ruptured aneurysm or any non-ruptured aneurysm on the same admission prior to enrollment.
5. SAH not caused by aneurysm rupture or aneurysm is identified to be traumatic, mycotic, blister or fusiform type by catheter Digital Subtraction Angiography (DSA).
6. Any intracranial stent placement or non-coil intra-aneurysmal device (i.e., stent- assisted coiling with Neuroform, Enterprise, LVIS, LVIS Jr, Barrel Stent, Pulse Rider, LUNA, Medina or a similar device) where the stent device is implanted to treat the ruptured aneurysm and / or antiplatelet therapy is needed.
7. Subject has remaining aneurysm(s) that are untreated and could reasonably be considered a possible alternate cause of the aSAH based on the observed bleeding pattern. Adequate treatment of these aneurysms by coiling embolization would result in the aneurysms no longer causing an exclusion. MRI may be used in some situations to determine that the associated aneurysms did not rupture based on lack of blood seen adjacent to the additional aneurysms.
8. Diagnosis of sepsis (systemic inflammatory response syndrome [SIRS] criteria plus the presence of known or suspected infection) or current documented active bacterial or viral infection prior to enrollment (Example: significant upper respiratory infection (URI), community-acquired pneumonia). A minor non-complicated community-acquired urinary tract infection (UTI) would not be an exclusion but should be treated promptly.
9. New parenchymal hemorrhage or new infarction larger the 15 milliliters in volume, or significant increased mass effect as seen on the post coiling pre-enrollment head CT when compared to baseline admission head CT. New hyperdensity on CT scan related to contrast staining is not an exclusion.
10. Subject developed SAH-induced cardiac stunning prior to enrollment, with an ejection fraction< 30%, or requiring intravenous medications for blood pressure maintenance.
11. Concurrent significant intracranial pathology identified prior to enrollment, including but not limited to, Moyamoya disease, high suspicion or documented CNS vasculitis, severe fibromuscular dysplasia, arteriovenous malformation, arteriovenous fistula, significant cervical or intracranial atherosclerotic stenotic disease (greater or equal to 70%), or malignant brain tumor.
12. Known seizure or epilepsy disorder (diagnosed prior to this aSAH diagnosis) where anti-epileptic medication was previously taken by the patient or have been recommended to be taken by the patient. Childhood seizures that have resolved and no longer require treatment are not part of this exclusion criteria.
13. Serious co-morbidities that could confound study results including but not limited to: Multiple Sclerosis, dementia, severe major depression, cancer likely to cause death in 2 years, multi-system organ failure, or any other conditions that could cause any degree of cognitive impairment.
14. Immunosuppression therapy including chronic corticosteroid usage.
15. Remote history of previous ruptured cerebral aneurysm.
16. History of gastrointestinal hemorrhage or major systemic hemorrhage within 30 days, hemoglobin less than 8 g/dL, international normalized ratio greater than or equal to1.5, severe liver impairment, creatinine greater than 2.0 mg/dL, or estimated glomerular filtration rate less than 60 ml/min.
17. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days.
18. Currently pregnant.
19. Contraindication for MRI.
20. No hydrocephalus requiring EVD or LP.
21. Known hypersensitivity to Deferiprone or to any of the excipients in the formulation.
22. If endovascular treatment of their aneurysm requires adjunctive antiplatelet treatment.
23. Uncontrollable hypertension (>180 systolic and/or >110 diastolic) that is not correctable prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Ferritin levels in cerebrospinal fluid | Day 10 from enrollment
  Concentration of ferritin in the cerebrospinal fluid

SECONDARY OUTCOMES:
Assess functional outcomes | 6 and 12 months from enrollment
  Measured by the Montreal Cognitive Assessment (MoCA) score
Change in hippocampus size | On admission and at 6 and 12 months
  The size of hippocampus will be matched to historic control subjects matched with age, gender and level of education and measured using high resolution MRI
Change in amygdala measured size | On admission and at 6 and 12 months
  The size of amygdala will be matched to historic control subjects matched with age, gender and level of education and measured using high resolution MRI
Change in the amount of iron deposition in the brain | On admission and at 6 and 12 months
  Calculated using Quantitative susceptibility mapping (QSM) Magnetic Resonance Imaging (MRI)
Indications of clinical vasospasm | During hospitalization, up to 4 weeks
  Assessed during hospitalization
Indications for delayed cerebral ischemia | During hospitalization, up to 4 weeks
  Assessed during hospitalization
Incidence of hydrocephalus requiring shut placement | During hospitalization, up to 4 weeks
  Assessed during hospitalization
Change in Modified Rankin Scale (mRS) score | At 6 weeks, and 6 and 12 months
  Documented at 6 weeks, and 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Hasan, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Univesity of Iowa Hospital and Clinics, Iowa City, Iowa
  - Duke University Health System, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van der Loo LE, Aquarius R, Teernstra O, Klijn K, Menovsky T, van Dijk JMC, Bartels R, Boogaarts HD. Iron chelators for acute stroke. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD009280. doi: 10.1002/14651858.CD009280.pub3. PMID 33236783

DOCUMENTS (1):
  • Informed Consent Form (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03754725/ICF_001.pdf